CLINICAL TRIAL: NCT02107079
Title: The Relative Bio-availability of Oral and Oromucosal Melatonin in Different Formulations in Healthy Human Volunteers. A Three-phased Cross-over Study.
Brief Title: The Relative Bio-availability of Oral and Oromucosal Melatonin in Different Formulations in Healthy Human Volunteers.
Acronym: Melaform
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Utrecht University (Other)
Responsible Party: Principal Investigator, Ingeborg Marianne van Geijlswijk, hospital pharmacist, Utrecht University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Melaform; 2011-003068-61 (EudraCT Number)
Record Dates: First submitted 2014-04-03; First posted 2014-04-08 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-04

CONDITIONS: Pharmacokinetics of Melatonin
Keywords: melatonin; bioavailability; pharmacokinetics
MeSH Terms: interventions — Melatonin

ARMS (3):
- melatonin 1 mg immediate release tablet (Active Comparator)
  Interventions: Drug: Melatonin
- melatonin 2,5mg immediate release capsule (Active Comparator)
  Interventions: Drug: Melatonin
- melatonin 0.1 mg oromucosal tablet (Active Comparator)
  Interventions: Drug: Melatonin

INTERVENTIONS:
Drug: Melatonin — swallowing 1 piece, collecting saliva afterwards
  Other Names: Melatonin 2,5 mg capsule (compounded by UMCU Pharnacy); Melatonin 1 mg tablet Thiopharma; Sleepzz 0.1 mg oromucosal tablet

SUMMARY:
The circadian rhythm, the sleep-wake cycle, is mainly regulated by melatonin. The synthesis of melatonin is stimulated by the absence of light, leading to peak serum levels before bedtime. In humans, this endogenous "signaling" neurohormone induces sleep. Exogenous melatonin can be beneficial in different sleep disturbances including delayed sleep phase insomnia, melatonin- deficiency-related insomnia (especially in elderly) and shift work sleep disorder. Melatonin is known for its low and variable bioavailability in humans due to a high first pass effect and variable pharmacokinetics and short half-life. In order to prevent exposure of patients with unnecessary high dosages of melatonin and in order to achieve a short Tmax and high bio-availability of melatonin, a proper formulation needs to be defined. This study, a three-phased cross-over study, aims to define a proper formulation for oral and oromucosal melatonin for the treatment of insomnia by investigating the Tmax and relative bioavailability derived from melatonin levels in salivary samples of healthy volunteers after administration of melatonin in different formulations: 2,5mg melatonin immediate release capsule (produced by Apotheek UMCU), 1mg melatonin immediate release tablet (produced by Tiofarma), low-dose 0.1mg melatonin original Sleepzz tablet (produced by Vemedia Manufacturing BV).

DETAILED DESCRIPTION:
The circadian rhythm, the sleep-wake cycle, is mainly regulated by melatonin. The synthesis of melatonin is stimulated by the absence of light, leading to peak serum levels before bedtime. In humans, this endogenous "signaling" neurohormone induces sleep.

Exogenous melatonin can be beneficial in different sleep disturbances including delayed sleep phase insomnia (Dahlitz et al. 1991, Regestein et al. 1995), melatonin- deficiency-related insomnia (especially in elderly) (Garfinkel 1995, Etzioni et al. 1995) and shift work sleep disorder (Folkard et al. 1993, Skene et al. 1996).

A randomized controlled trial of van Geijlswijk et al. (van Geijlswijk 2010) showed that no relationship could be demonstrated between melatonin dose (0.05-0.15 mg/kg) and shift of sleep onset time (SOT), shortening of sleep onset latency (SOL) and shift of dim light melatonin (DLMO). On the other hand, the timing of melatonin administration did have a clinically and statistically significant effect on all three parameters. Timing of melatonin administration in relation to baseline DLMO determines the phase advance, as can be measured by the shift of DLMO and SOT to an earlier time in the evening, resulting also in a shorter SOL. Melatonin must be administered in a closely defined time-slot before endogenous DLMO and before bedtime. The phase advance occurs when melatonin is administered 1-2 hours before DLMO and bedtime (van Geijlswijk et al. 2010). This trial demonstrated that low dosage of melatonin (0.05mg/kg) is effective in children when given at least 1-2 hours before the individual DLMO and the desired bedtime. This means that the release of melatonin from any pharmaceutical formulation should occur fast enough in order to achieve predictive high levels within the desired time-slot before the occurrence of (baseline) DLMO to induce a phase advance. These high maximum serum levels shortly after administration (Tmax) means the release rate of melatonin from the formulation needs to be as fast as possible and the bioavailability needs to be as high as possible.

Melatonin is known for its low and variable bioavailability in humans due to a high first pass effect and variable pharmacokinetics and short half-life. In order to prevent exposure of patients with unnecessary high dosages of melatonin and in order to achieve a short Tmax and high bio-availability of melatonin, a proper formulation needs to be defined. Thereby, the bioavailability must be made less variable in order to understand the biologic effects of melatonin (Di 1997).

Aim/objective. This study, a three-phased cross-over study, aims to define a proper formulation for oral and oromucosal melatonin for the treatment of insomnia by investigating the Tmax and relative bioavailability derived from melatonin levels in salivary samples of healthy volunteers after administration of melatonin in different formulations: 2,5mg melatonin immediate release capsule (produced by Apotheek UMCU), 1mg melatonin immediate release tablet (produced by Tiofarma), low-dose 0.1mg melatonin original Sleepzz tablet (produced by Vemedia Manufacturing BV).

Study-design. Three-phased cross-overstudy. Study-population. The study population will consist of 10 healthy volunteers (male) aged 18 to 35 years old without insomnia. They will be recruited in the Netherlands. Intervention. The intervention starts between 10:00 and 11:00 am when the participant flushes his mouth with water, waits 15 minutes and starts to chew on a cotton plug during 1 minute. Directly after that the participant will administer one of the IMP's according to the instructions. The tablet and capsule will be swallowed. The sublingual tablet will be administered sublingual. 10 minutes after administration the subjects will drink one glass of water and subsequently try to swallow as much liquid (including saliva), in order to prevent contamination of the saliva sample with the remaining exogenous melatonin. At 15 minutes, 30 min, 1 hour, 1.5 hour, 2 hours and 3 hours after oral administration the participant will chew on new cotton plugs during 1 minute. After administration of the sublingual tablet saliva samples will be collected at 25 minutes, 40 minutes, 60 minutes, 1.5 hour, 2 hours and 3 hours after sublingual administration. 15 minutes before each sampling the subject will flush his mouth with water. The cotton plugs with salivary will be preserved in a test-tube in the freezer and will be analyzed by Ziekenhuis Gelderse Vallei.

Main study endpoint: the Tmax and relative bioavailability of oral and oromucosal melatonin derived from melatonin levels in salivary samples of healthy volunteers.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

This study will burden the participants in a small extent. As mentioned before, melatonin is well tolerated and is not reported to have a hangover effect. Its rarely occurring side effects include fatigue, dizziness, nausea, mild drowsiness, hypothermia and headache (Wagner 1998, Waldhauser 1990, Dahlitz 1991, Garfinkel 1995, Dollins 1994). Besides that, the participants will be asked to perform simple actions during 3 intervention days for only 3 hours.

The low dose 0.1mg melatonin original Sleepzz table is available without prescription in drugstores in the Netherlands. The tablet will also contain low dosage of melatonin, respectively 1mg and the capsule will contain regular dose of melatonin (2,5mg). These dosages are safe for adults and children. A few reports have been published on the consequences of long-term treatment with melatonin in humans. (Severe) adverse events were not described in these reports. (Van Geijlswijk 2011, Jan et al. 1996, Jan et al. 1994, Gilberg et al. 1997, Smits et al. 2001, Arendt 2000).

ELIGIBILITY:
Inclusion Criteria:

* Volunteers (male) aged from 18 to 35 years old without insomnia.

Exclusion Criteria:

* Lactose intolerance.
* Hepatic disease
* Kidney disease
* Auto-immune disease
* Depression
* Neurological disorders
* Oromucosal diseases.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2012-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Melatonin concentration (ng/ml) in saliva | At 15 min, 30 min, 1 hour, 1.5 hour, 2 hours, 3 hours (tablet; capsule); at 25 minutes, 40 minutes, 60 minutes, 1.5 hour, 2 hours and 3 hours (sublingual tablet )

CONTACTS AND LOCATIONS:
Locations (1):
- Pharmacy department of faculty of veterinary medicine Utrecht University, Utrecht, Utrecht, Netherlands

REFERENCES:
- See also: CCMO protocol — https://www.toetsingonline.nl/to/ccmo_search.nsf/fABRpop?readform&unids=C1257BA2002CC066C125799F0031679F